CLINICAL TRIAL: NCT01259349
Title: Standard Coaxial Microincision Cataract Surgery Versus Coaxial Microincision Cataract Surgery Using 1% Ultrasound in Immature Senile Cataract :a Corneal Endothelium Study
Brief Title: Effect of Minimising Ultrasound Power to 1% During Cataract Surgery on Corneal Endothelium.
Acronym: OCTOPUS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Ram Manohar Lohia Hospital (Other Government)
Responsible Party: Dr. Taru Dewan, Dr. Ram Manohar Lohia Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RMLH-002-EYE
Record Dates: First submitted 2010-12-06; First posted 2010-12-14 (Estimated); Last update posted 2010-12-15 (Estimated); Status verified 2010-11

CONDITIONS: Cataract
Keywords: cataract,; phacoemulsification,; one percent ultrasound; endothelial cell density
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- one percent ultrasound (Experimental): Co-axial MICS shall be performed in cases allocated to this arm .The ultrasound power shall be kept at one percent during the surgery.A note of effective phacotime,volume of fluid aspirated and any intraoperative complications shall be made.
  Interventions: Procedure: one percent ultrasound power in CMICS
- 40 percent ultrasound (Active Comparator): Co-axial MICS shall be performed in cases allocated to this arm .The ultrasound power shall be kept at 40 percent during the surgery.A note of effective phacotime,volume of fluid aspirated and any intraoperative complications shall be made.
  Interventions: Procedure: 40 percent ultrasound power in CMICS

INTERVENTIONS:
Procedure: one percent ultrasound power in CMICS — Co-axial MICS shall be performed in cases allocated to this arm .The ultrasound power shall be kept at one percent during the surgery.A note of effective phacotime,volume of fluid aspirated and any intraoperative complications shall be made.
  Other Names: OCTOPUS
  Arms: one percent ultrasound
Procedure: 40 percent ultrasound power in CMICS — Co-axial MICS shall be performed in cases allocated to this arm .The ultrasound power shall be kept at 40 percent during the surgery.A note of effective phacotime,volume of fluid aspirated and any intraoperative complications shall be made.
  Other Names: standard CMICS
  Arms: 40 percent ultrasound

SUMMARY:
Coaxial microincision cataract surgery using 1% ultrasound is not inferior to standard coaxial microincision cataract surgery in patients of grade 0.1-6.0 immature senile cataract in terms of corneal endothelial safety.

DETAILED DESCRIPTION:
Corneal endothelial damage and posterior capsular rupture are two most undesirable complications of cataract surgery, infact significant loss of endothelium can lead to corneal decompensation and loss of corneal clarity. However, some degree of endothelial cell loss is inevitable after any cataract surgery. A loss of 3.2%-23.2% has been shown in various studies since 1967. It is well known that during cataract surgery many different factors can generate endothelial damages, these include the impact of the nuclear fragments, the turbulence generated in anterior chamber and the volume of liquid. It is also related to the amount of ultrasonic energy used and the subsequent temperature rise, the contact with surgical instruments and the IOL during implantation. It also depends on the release of free radicals the length and features of incision,the surgical technique used . The risk of endothelial cell density loss is further enhanced when surgeons have to deal with high density cataract, shallow anterior chamber and old age.

Since the time Kelman introduced his technique of phacoemulsification, there has been constant and conscious effort on the part of phaco surgeons to reduce their phaco time by bringing some alteration or innovation in their personal technique or introducing new technologies for the procedure of phacoemulsification. Development of Laser emulsifier, SONAAR machines, introduction of cold phaco with modulations of ultrasound in the form of pulse, micropulse and bursts were achievements towards attaining this end and goal.

Coaxial microphacoemulsification is the standard phacoemulsification technique being practised globally for cataract extraction and on many occasions we intentionally do not use the phaco power either at all or fully as per the pre set limit. In fact the use of efficient fluidic controls and a chopper minimizes the use of phaco energy. If we could assess a zero/minimal ultrasound technique in a scientific setting we might achieve the desired goal without resorting to major modifications of instrumentation and machine. Coaxial MICS fully utilizes the advantages of small incision and provides the most comfortable platform for the surgeons using conventional phacoemulsification.

We imagined that most ideal setting would be introducing zero phaco power in the anterior chamber for emulsifying the nucleus as has been done already in case of Aqualase using warm fluid based system and Howard Fines new technique of mechanically emulsifying the lens with rotators(under investigation). For that we undertook a pilot study in 10 patients and performed coaxial microincision phacoemulsification, introducing the ultrasound power in incremental fashion during the surgery in each of the 10 patients till we could achieve the adequate aspiration of fluid and fragments .

At zero power the phacotip and tubing experienced repeated blockages with associated prolongation of surgical time,thus increment to one percent was made during the same sitting. To our surprise, the very first step of introducing 1% ultrasound power made all the difference.No further increments were required as all techniques of nuclear management and lens aspiration were conveniently possible at this setting.

The procedure of aspiration of fragments was smooth and continuous, it also caused a reduction in the surgical time in comparison to zero power phaco.The cases revealed less corneal endothelial trauma in comparison to conventional phacoemulsification using higher power settings. The most surprising observation was that we could dissemble the nucleus with any known technique of nucleus fragmentation(stop and chop, divide and conquer, phaco-chop) in almost all grades of cataracts .Possibly that high vaccum 300-350 is responsible for this nuclear fragmentation and not only the cavitational effects of ultrasound power.

Keeping all the other parameters uniform we wish to design an RCT to study the effect of eliminating phaco power. With this in view,this study compares the endothelial status in addition to various complications and visual outcome following standard coaxial microincision cataract surgery and coaxial microincision cataract surgery using 1% ultrasound.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of >40yrs will be included in the study.
2. Grade 0.1-6.0 (LOCS III grading) of senile cataract.

Exclusion Criteria:

1. Patients with pre-operative endothelial cell density count less than 1500cells/mm2.
2. All eye pathologies that can compromise the visual recovery.
3. Eyes with any kind of corneal dystrophy or corneal scars preventing visualisation of cataract for reliable grading.
4. Raised intraocular pressure (> 21 mmHg).
5. Previous intraocular surgery.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
change in endothelial cell count from baseline over time | 1 day,1week,months 1,3,6,9,12
  Noncontact specular microscope (EM - 3000; TOMEY: VERSION 2A/OJ) will be used to calculate the endothelial cell density, coefficient of variation of cell size, percentage of hexagonal cells and corneal thickness before surgery and 1day, 1 week, 1, 3, 6, 9 and 12 months visits after surgery. 3 endothelial cell photographs will be taken at each visit and the mean cell count of three photographs will be calculated. Counts will be performed by an observer blinded to which procedure the patient had undergone. Endothelial cell loss will be calculated as a percentage of pre operative cell density

SECONDARY OUTCOMES:
change in Intraocular pressure from baseline | 1day,1week,months1,3,6,9,12
  Intraocular pressure will be measured using applanation tonometer.
visual acuity | 1 month
  snellens visual acuity will be converted to Logmar scale and recorded with and without spectacle correction
posterior capsular rupture | day 0 of surgery
  any incidence of posterior capsular rupture during surgery would be noted

CONTACTS AND LOCATIONS:
Overall Officials: Taru Dewan, MS FRCSEd, Principal Investigator — Dr. R.M.L.Hospital,New Delhi,India
Locations (1):
- Dr. R.M.L.Hospital,, New Delhi, National Capital Territory of Delhi, India